CLINICAL TRIAL: NCT03500939
Title: Penumbral Rescue by Normobaric O=O Administration in Patients With Ischemic Stroke and Target Mismatch ProFile: A Phase II Proof-of-Concept Trial
Brief Title: Penumbral Rescue by Normobaric O2 Administration in Patients With Ischemic Stroke and Target Mismatch ProFile
Acronym: PROOF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Coordination Centre for Clinical trials (KKS), 69120 Heidelberg, Germany (Unknown); European Clinical Research Infrastructure Network (ECRIN), 10559 Berlin, Germany (Unknown); CORE IMAGING LABORATORY: Eppdata GmbH, 22529 Hamburg, Germany (Unknown); CORE BIOMARKER LABORATORY: Fundatio Hospital Universitari Vall d'Hebron, 08035 Barcelona, Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROOF; 2017-001355-31 (EudraCT Number)
Record Dates: First submitted 2018-03-27; First posted 2018-04-18 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normobaric hyperoxygenation + standard of care (Experimental): Normobaric hyperoxygenation (NBHO), i.e. inhalation of 100% oxygen at high flow (≥ 40 L/min) via a sealed non-rebreather face-mask with reservoir, or in case of intubation/ventilation for (study-independent) TBY, ventilation with an inspiratory oxygen fraction (FiO2) of 1.0. NBHO is started within 3 hours of stroke symptom onset (witnessed or last seen well) and within 20 minutes after end of baseline brain imaging and applied until the end of TBY procedure (defined by removal of guide catheter from sheath) or, in case TBY is not attempted, 4 hours after start of study treatment.
  Interventions: Drug: Medical oxygen; Other: Standard of care
- standard of care alone (Active Comparator): standard of care alone; oxygen supplementation if SpO2 ≤ 94% at 2 to 4 L/min via nasal cannula according to guidelines of the European Stroke Organisation (ESO), or in case of TBY-related intubation/ventilation, ventilation with an initial FiO2 of 0.3 to be gradually increased if SpO2 ≤ 94%.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Medical oxygen — inhalation of 100% oxygen at high flow via a sealed non-rebreather face-mask with reservoir
  Arms: Normobaric hyperoxygenation + standard of care
Other: Standard of care — e.g. thrombectomy, thrombolysis

SUMMARY:
The main objective of the PROOF trial is to investigate efficacy and safety of normobaric hyperoxygenation (NBHO) as a neuroprotective treatment in patients with acute ischemic stroke due to large vessel occlusion likely to receive endovascular mechanical thrombectomy (TBY) in a randomized controlled clinical phase IIb trial.

DETAILED DESCRIPTION:
http://www.proof-trial.eu/

European Union's Horizon 2020 research and innovation programme grant 733379 (2016): Euro 5.8 Mio

ELIGIBILITY:
Inclusion Criteria

* Age: >= 18 years
* Acute anterior circulation ischemic stroke due to an LVO on CT or MR angiography, i.e. either terminal ICA with M1/carotid-T, proximal M1, distal M1 (distal to perforating branches), or M2/3 segment(s)
* If TBY is likely to be conducted* (*However, neither TBY nor IVT are a prerequisite for inclusion; patients not receiving TBY or IVT or both can be enrolled. Clinical treatment decisions should not delay study enrollment).
* NIHSS score of ≥ 6 at screening
* ASPECTS of 7-10 on NCCT or 6-10 on DWI-MRI
* CT or MR perfusion (whole-brain or minimal coverage ≥ 75 mm) prior to NBHO
* NBHO can be initiated within 6 hours of symptom onset (witnessed or last seen well) and within 30 minutes after last image of baseline brain imaging
* Pre-stroke mRS of 0 or 1
* Breastfeeding women must stop breastfeeding after randomization
* Own written informed consent is not obtained prior to study inclusion but has to be gained as soon as possible. Patients who are able to give consent will be informed about trial participation orally and may consent to or decline participation. Patients unable to give consent will be enrolled through a deferred consent procedure.

Exclusion Criteria

Neurological:

* TBY procedure initiated (groin puncture) prior to randomization
* Rapid major improvement in neurological status prior to randomization
* Any condition which precludes obtaining an accurate baseline NIHSS or outcome assessment (e.g. seizures, dementia, psychiatric or neuromuscular disease)
* Intracranial hemorrhage (except of cerebral microbleeds), intracranial tumor (except small meningioma), and/or intracranial arteriovenous malformation
* Intracranial aneurysm or prior stent implantation in the vascular territory (upstream and downstream) affected by qualifying LVO
* Suspected complete CCA occlusion, aortic dissection, cerebral vasculitis, septic embolism, or bacterial endocarditis
* Acute bilateral stroke or stroke in multiple vascular territories (except of clinically silent micro-lesions)

Respiratory:

* Known history of chronic pulmonary disease (e.g. COPD, pulmonary fibrosis, alveolitis or pneumonitis)
* Prior to enrolment, > 2 L/min oxygen required to maintain peripheral oxygen saturation ≥ 95%
* Acute respiratory distress that may, in the clinical judgment of the investigator, interfere with the study intervention
* Acute pneumonia, alveolitis or pneumonitis of viral, bacterial, fungal or any other etiology

Other:

* Clinical suspicion of acute myocardial infarction (e.g. acute chest pain)
* Baseline blood glucose of < 50 mg/dL (2.78 mmol) or > 400 mg/dL (22.20 mmol)
* Body temperature ≥ 38.0°C at screening
* History of severe allergy (more than rash) to contrast medium
* Current treatment with nitrofurantoin or amiodaron, paraquat poisoning, or history of treatment with bleomycin
* Pregnancy at screening, to be excluded (β-HCG in serum or urine) in all women ≤ 55 years except if surgically sterile; in women >55 years pregnancy must be excluded only in case of increased probability e.g. due to in-vitro fertilization
* Any co-existing or terminal disease (except qualifying stroke) with anticipated life expectancy of less than 6 months
* Any pre-existing condition that may, in the clinical judgment of the investigator, not allow safe participation in the study (e.g. alcohol or substance abuse, co-existing disease)
* Participation in another interventional (drug or device) study within the last four weeks
* Prior participation in the PROOF trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
ischemic core growth from baseline to 24 hours | from baseline to 24 (22 to 36) hours
  difference in ischemic core volume (in mL) from baseline to 24 hours; intention-to-treat (ITT) analysis

SECONDARY OUTCOMES:
change in National Institutes of Health Stroke Scale (NIHSS) score from baseline to 24 hours | from baseline to 24 ± 6 hours
  key secondary endpoint; the NIHSS is a stroke severity score that is composed of 11 items; range from 0 to 41, higher values indicate more severe deficits
survival | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; survival to be assessed at visit 6 (V6, day 5), and V7 (day 90)
National Institutes of Health Stroke Scale score (NIHSS) | 20 ± 10 minutes, 4 hours ± 15 minutes, 24 ± 6 hours, 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; NIHSS to be assessed at visit 2 (V2, 20 minutes), V4 (end of study treatment), V5 (24 hours), V6 (day 5), and V7 (day 90); the NIHSS is a stroke severity score composed of 11 items (range from 0 to 41, higher values indicate more severe deficits)
modified Rankin Scale score (mRS) | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; mRS to be assessed at visit 6 (V6, day 5), and V7 (day 90); the mRs is an ordinal disability score of 7 categories (0 = no symptoms to 5 = severe disability, and 6 = death)
Barthel Index (BI) | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; BI to be assessed at visit 6 (V6, day 5), and V7 (day 90)
Montreal Cognitive Assessment (MoCA) | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; MoCA to be assessed at visit 7 (day 90)
Stroke Impact Scale 16 (SIS-16) | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; SIS-16 to be assessed at visit 7 (day 90); the SIS-16 is a 16-item physical dimension instrument for measuring the physical aspects of stroke recovery (items are rated on a 1 to 5 scale; 5 = not difficult at all, 1 = could not do at all)
EuroQoL Questionnaire (EQ-5D-5L) | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; EQ-5D-5L to be assessed at visit 7 (day 90)
Montgomery-Åsberg Depression Rating Scale (MADRS) | 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; MADRS to be assessed at visit 7 (day 90); the MADRS is a 10-item depression rating test that uses a 0 to 6 severity scale (higher scores indicate increasing depressive symptoms)
partial pressure of oxygen in the arterial blood (PaO2) | 90 ± 30 minutes, 24 ± 6 hours after randomization
  secondary clinical efficacy endpoint; PaO2 to be assessed at visit 3 (90 minutes after start of study treatment), and V5 (24 hours)
length of ICU stay | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; length of ICU stay to be assessed at visit 6 (V6, day 5), and V7 (day 90); ICU is defined as a ward with capacity for mechanical ventilation and/or continuous monitoring of vital parameters (including stroke units)
length of hospital stay | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; length of hospital stay to be assessed at visit 6 (V6, day 5), and V7 (day 90)
duration of ventilation | 5 ± 2 days, 90 ± 10 days after randomization
  secondary clinical efficacy endpoint; duration of ventilation to be assessed at visit 6 (V6, day 5), and V7 (day 90)
all-cause death | 5 ± 2 days, 90 ± 10 days after randomization
  clinical safety endpoint; to be assessed at visit 6 (V6, day 5), and V7 (day 90)
stroke related death | 5 ± 2 days, 90 ± 10 days after randomization
  clinical safety endpoint; to be assessed at visit 6 (V6, day 5), and V7 (day 90)
symptomatic intracranial hemorrhage | 5 ± 2 days after randomization or discharge
  clinical safety endpoint; per ECASS III definition and per Heidelberg bleeding classification
vital signs | 90 ± 10 days after randomization
  clinical safety endpoint; systolic and diastolic blood pressure, heart and respiratory rate, peripheral capillary oxygen saturation (SpO2)
12-lead electrocardiogram (ECG) | 24 ± 6 hours after randomization
  clinical safety endpoint
safety laboratory | 5 ± 2 days after randomization or discharge
  clinical safety endpoint; blood count, clinical chemistry, coagulation
concomitant invasive procedures | 90 ± 10 days after randomization
  clinical safety endpoint; e.g. intravenous/intra-arterial thrombolysis, thrombectomy, stenting, carotid surgery, decompressive hemicraniectomy, cardioversion, patent foramen ovale (PFO) closure
relative changes in ischemic core volume (in %) from baseline to 24 hours | from baseline to 24 (22 to 36) hours
  secondary imaging efficacy endpoint
absolute and relative ischemic core change from baseline to 24 hours using cerebral blood flow (CBF) < 30% for ischemic core estimation at baseline in all patients | from baseline to 24 (22 to 36) hours
  secondary imaging efficacy endpoint; independent of imaging modality
penumbral salvage from baseline to 24 hours | from baseline to 24 (22 to 36) hours
  secondary imaging efficacy endpoint
TICI (Thrombolysis in Cerebral Infarction perfusion scale grade) | 4 hours ± 15 minutes
  secondary imaging efficacy endpoint; in patients who underwent mechanical thrombectomy (TBY)
revascularization on 24-hour follow-up imaging | 24 (22 to 36) hours
  secondary imaging efficacy endpoint
new microbleeds on 24-hour follow-up MRI (vs. baseline T2*weighted MRI) | 24 (22 to 36) hours
  imaging safety endpoints; only possible in patients who had MRI at baseline as well as at 24 hours
any intracranial hemorrhage on 24-hour follow-up imaging | 24 (22 to 36) hours
  imaging safety endpoints
peri-interventional occurrence of vasospasms | 4 hours ± 15 minutes
  imaging safety endpoints; in patients who underwent mechanical thrombectomy (TBY)
ischemic lesions in new territories on 24-hour follow-up imaging | 24 (22 to 36) hours
  imaging safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Sven Poli, MD, Principal Investigator — University Hospital Tübingen
Locations (22):
- Belgium (4):
  - UZ Gent, Ghent
  - AZ Groeninge Kortrijk, Kortrijk
  - KU Leuven, Leuven
  - CHU de Liège, Liernu
- Helsinki University Hospital, Helsinki, Finland
- France (5):
  - CHU de Grenoble, Grendelbruch
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - Centre Hospitalier Saint Anne de Paris, Paris
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
- Germany (9):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Gießen, Giessen
  - Universitätsklinikum Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - Ludwig-Maximilians-Universität München, München
  - St. Lukas Klinik, Solingen
  - University Hospital Tuebingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Spain (3):
  - Fundacio Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - HCU Valladolid, Valladolid

REFERENCES:
- [Derived] Poli S, Mbroh J, Baron JC, Singhal AB, Strbian D, Molina C, Lemmens R, Turc G, Mikulik R, Michel P, Tatlisumak T, Audebert HJ, Dichgans M, Veltkamp R, Husing J, Graessner H, Fiehler J, Montaner J, Adeyemi AK, Althaus K, Arenillas JF, Bender B, Benedikt F, Broocks G, Burghaus I, Cardona P, Deb-Chatterji M, Cvikova M, Defreyne L, De Herdt V, Detante O, Ernemann U, Flottmann F, Garcia Guillamon L, Glauch M, Gomez-Exposito A, Gory B, Sylvie Grand S, Harsany M, Hauser TK, Heck O, Hemelsoet D, Hennersdorf F, Hoppe J, Kalmbach P, Kellert L, Kohrmann M, Kowarik M, Lara-Rodriguez B, Legris L, Lindig T, Luntz S, Lusk J, Mac Grory B, Manger A, Martinez-Majander N, Mengel A, Meyne J, Muller S, Mundiyanapurath S, Naggara O, Nedeltchev K, Nguyen TN, Nilsson MA, Obadia M, Poli K, Purrucker JC, Raty S, Richard S, Richter H, Schilte C, Schlemm E, Stohr L, Stolte B, Sykora M, Thomalla G, Tomppo L, van Horn N, Zeller J, Ziemann U, Zuern CS, Hartig F, Tuennerhoff J; PROOF investigators. Penumbral Rescue by normobaric O = O administration in patients with ischemic stroke and target mismatch proFile (PROOF): Study protocol of a phase IIb trial. Int J Stroke. 2024 Jan;19(1):120-126. doi: 10.1177/17474930231185275. Epub 2023 Aug 18. PMID 37515459
- See also: Related Info — http://www.proof-trial.eu/